CLINICAL TRIAL: NCT05185141
Title: Assessing Respiratory Variation of Carotid Doppler Peak Velocity (CDPV) for Non-invasive Prediction of Fluid Responsiveness During Abdominal Surgery: a Prospective Observational Trial
Brief Title: Respiratory Variation of Carotid Doppler Peak Velocity (CDPV) for Non-invasive Prediction of Fluid Responsiveness
Status: Recruiting | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Johannes M Wirkus, MD, Principal Investigator Johannes Wirkus, M.D., Johannes Gutenberg University Mainz
Other Study IDs: 21-02546
Record Dates: First submitted 2021-12-20; First posted 2022-01-11 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Hemodynamic Instability
Keywords: Fluid Responsiveness; Hemodynamic Monitoring; Carotid Doppler Peak Velocity; Pulse Pressure Variation; Fluid Challenge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess respiratory variation of carotid doppler peak velocity (∆CDPV) for prediction of fluid responsiveness during major abdominal surgery.

DETAILED DESCRIPTION:
Investigating hemodynamic parameters in a group of 19 ICU-patients with septic shock, respiratory variation of carotid doppler peak velocity (∆CDPV) has been shown to be able to predict fluid responsiveness. For patients receiving so called lung protective ventilation with a tidal volume of 6ml/kg ∆CDPV was superior for prediction of fluid responsiveness when compared to other well established parameters such as pulse pressure variation (∆PP).

Likewise in another study ∆CDPV has been shown to be superior to stroke volume variation (∆SV) for prediction of fluid responsiveness in patients with septic shock when ventilated with a tidal volume of ≥8ml/ kg.

All in all respiratory variation of carotid doppler peak velocity (∆CDPV) seems to be a promising parameter for prediction of fluid responsiveness (Yao et al., BMC Anesthesiology 2018). However, so far clinical studies have been conducted only under a small number of patients mainly in the intensive care unit and/ or under highly specific conditions (e.g. cardiac surgery).

If ∆CDPV is able to predict fluid responsiveness with high accuracy intraoperatively remains unknown. The investigators are therefore conducting this prospective monocentric observational trial to evaluate the performance of ∆CDPV during major abdominal surgery and compare it to validated fluid responsiveness monitoring parameters ∆PP and corrected flow time (fTc).

Following IRB-approval and written informed consent 84 patients scheduled for major abdominal surgery will be enrolled in the study. Stroke volume will be monitored by Esophageal Doppler Monitoring (CardioQ-ODM®, Deltex Medical Ltd, Chichester, UK). In case of hypovolemia a fluid bolus of 7 ml/kg ideal body weight will be administered at the discretion of the attending anesthesiologist. Respiratory variation of carotid doppler peak velocity (∆CDPV) will be monitored before and 1 minute after completion of each fluid bolus using an ultrasound device with a common linear array transducer (Philips ClearVue 350, Philips Medizin Systeme GmbH, Boeblingen, Germany).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* written informed consent
* scheduled major abdominal surgery

Exclusion Criteria:

* Age <18 or >80 years
* pregnancy
* SIRS or sepsis
* any kind of cardiac arrhythmia
* known valve disease
* known heart failure
* any kind of known carotid stenosis
* carotid doppler peak velocity >182 cm/s before baseline measurement (expected stenosis)
* missing indication for invasive arterial blood pressure monitoring (IBP) not related to the study
* peripheral artery disease (PAD)
* BMI > 35 kg/m2
* intraabdominal hypertension
* ASA-PSC of 4
* severe lung disease (e.g. COPD grade 3, fibrosis)
* esophageal disease of any kind
* participation in another clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only patients scheduled for major abdominal surgery with an expected high intraoperative fluid turnover will be eligble for the study. Patients with any kind of crdiac arrhythmia, valve diseases, heart failure or carotid stenosis will be excluded from the study to avoid measurement errors and bias for the hemodynamic parameters such as pulse pressure variation, stroke volume and carotid doppler peak velocity.
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in stroke volume following a fluid bolus. | Immediately before and 1 minute after completion of each fluid bolus.
  A rise in stroke volume of ≥10% following a fluid bolus of 7ml/kg Ideal Body Weight is considered to reflect fluid responsiveness. Measurements will be assessed through esophageal doppler monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Gunther J Pestel, M.D., Ph.D., Study Chair — Johannes Gutenberg University Medical Center, Dpt. of Anesthesiology; Kimiko Fukui-Dunkel, M.D., Ph.D., Study Director — Johannes Gutenberg University Medical Center, Dpt. of Anesthesiology
Locations (1):
- Department of Anesthesiology, Johannes-Gutenberg University Medical Center, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Background] Ibarra-Estrada MA, Lopez-Pulgarin JA, Mijangos-Mendez JC, Diaz-Gomez JL, Aguirre-Avalos G. Respiratory variation in carotid peak systolic velocity predicts volume responsiveness in mechanically ventilated patients with septic shock: a prospective cohort study. Crit Ultrasound J. 2015 Dec;7(1):29. doi: 10.1186/s13089-015-0029-1. Epub 2015 Jun 26. PMID 26123610
- [Background] Lu N, Xi X, Jiang L, Yang D, Yin K. Exploring the best predictors of fluid responsiveness in patients with septic shock. Am J Emerg Med. 2017 Sep;35(9):1258-1261. doi: 10.1016/j.ajem.2017.03.052. Epub 2017 Mar 22. PMID 28363617
- [Background] Yao B, Liu JY, Sun YB. Respiratory variation in peripheral arterial blood flow peak velocity to predict fluid responsiveness in mechanically ventilated patients: a systematic review and meta-analysis. BMC Anesthesiol. 2018 Nov 13;18(1):168. doi: 10.1186/s12871-018-0635-0. PMID 30424730